CLINICAL TRIAL: NCT00006504
Title: Flavonoids and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 945; R03HL065727 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Myocardial Infarction; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Stroke; Myocardial Infarction; Coronary Disease

SUMMARY:
To determine the association between flavonoids intake and the prevention of incident cardiovascular disease (CVD).

DETAILED DESCRIPTION:
BACKGROUND:

Basic science, clinical observation, and epidemiologic studies have all contributed to an emerging body of evidence on the potential role of flavonoids, a group of polyphenolic compounds with antioxidant properties, in the prevention of cardiovascular disease. However, the few existing studies on flavonoids or its food sources have provided inconsistent results, usually focusing on the primary prevention of coronary heart disease mortality. The study used the small grant mechanism (R03) to analyze previously collected data.

DESIGN NARRATIVE:

The investigators examined whether flavonoid intake was associated with the risk of incident CVD, and whether specific food sources of flavonoids--including tea, onions, apples, red wine, and other foods--were associated with the risk of incident CVD. The investigators processed and analyzed previously collected data of 39,876 middle-aged and older women free of CVD; the Women's Antioxidant Cardiovascular Study (WACS), a prospective study of 8,171 middle-aged and older women with pre-existing CVD or more than three coronary risk factors; the Normative Aging Study (NAS), a prospective study of 2,280 middle-aged and older men; and the Boston Area Health Study (BAHS), a case-control study of first nonfatal myocardial infarction in men and women aged less than 76 years. Using data from semiquantitative food frequency questionnaires administered in each study, the investigators determined individual intake of flavonoids and its food sources. Unlike previous studies, they examined flavonoids in relation to both the primary and secondary prevention of incident cardiovascular disease (CVD), consisting of confirmed cases of nonfatal myocardial infarction (Ml), nonfatal stroke, revascularization procedures, and CVD death.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Sesso — Brigham and Women's Hospital

REFERENCES:
- [Background] Sesso HD, Liu S, Gaziano JM, Buring JE. Dietary lycopene, tomato-based food products and cardiovascular disease in women. J Nutr. 2003 Jul;133(7):2336-41. doi: 10.1093/jn/133.7.2336. PMID 12840203
- [Background] Sesso HD, Gaziano JM, Liu S, Buring JE. Flavonoid intake and the risk of cardiovascular disease in women. Am J Clin Nutr. 2003 Jun;77(6):1400-8. doi: 10.1093/ajcn/77.6.1400. PMID 12791616